CLINICAL TRIAL: NCT03376282
Title: The Effect of Hyperbaric Oxygen Therapy on Kidney Function, Perfusion, Fibrosis and Proteinuria in Diabetic Patients With Diabetic Kidney Disease
Brief Title: Hyperbaric Oxygen Therapy for Renal Regeneration in Diabetic Nephropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in recruiting.
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shay Efrati, Head of HyperBaric center assaf-Harofhe MC, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 84-15
Record Dates: First submitted 2016-03-25; First posted 2017-12-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Renal Failure
Keywords: HBO; kidney functions; markers
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBOT treatment (Other): HBOT treatment: 60 daily sessions, 5 days/week, 120 minutes each, 100% oxygen at 2ATA.
  Interventions: Other: Hyperbaric Oxygen oxygen therapy (HBOT)
- Standard treatment (No Intervention): follow up with the standard recommended treatment

INTERVENTIONS:
Other: Hyperbaric Oxygen oxygen therapy (HBOT) — 60 daily sessions, 5 days/week, 120 minutes each, 100% oxygen at 2ATA.
  Arms: HBOT treatment

SUMMARY:
Diabetes kidney disease is a leading cause for end stage renal disease in the western world. To date no treatment that can reverse renal damage exists.

Chronic hypoxia is one of the major key insults affecting the diabetic kidney, and many of the new treatments under study focus on it's consequences, but no treatment can improve the hypoxia as both increased renal perfusion and decreased renal perfusion may be associated with it's worsening. Hyperbaric oxygen therapy (HBOT) can improve renal hypoxia by increasing partial pressure of dissolved (non-hemoglobin-bound) oxygen without affecting it's demand. HBOT also recruits tissue and peripheral progenitors and supplies the optimal environment crucial for their proliferation and for tissue repair. Hyperbaric oxygen treatment was known for years as an effective treatment for diabetic ulcers. Recent trials have shown great impact on brain lesions (in diabetic and non-diabetic patients) it is now the time to evaluate the effect of HBOT on the diabetic kidney.

DETAILED DESCRIPTION:
Scientific background

Diabetic Kidney Disease (DKD):

The kidneys, which are an important target for diabetic induced damage, contribute a lot to this burden. Diabetic nephropathy (DN) is the most common cause of end-stage kidney disease worldwide, associated with increased morbidity and mortality in patients with diabetes.

The pathogenesis of DKD is relatively established, less progress however have been achieved in the effort to heal the diabetic kidney. Current therapies aimed to control blood glucose levels and blood pressure, and in particular, inhibition of the RAS in order to prevent the development of albuminuria and progression of DKD. Many new therapies emerging recently have offered some potential, but yet none of them had proven effect on the renal progression.

While TGF beta1, MAPK, HIF, VEGF and others have stand in the focus of trials, and drugs that control each of these mediators were offered as the drug that will "make the change" these mediators are probably not the key insult.

Oxygen and the kidney

The kidneys consist of only 1% of the body weight, but consume more than 10% of its total oxygen consumption. Eighty percent of the oxygen is being consumed by the Na/K ATPase in the proximal tubule.

For most organs tissue oxygen tension is determined by the balance between the blood flow and tissue oxygen consumption. However, the kidneys do not fall under such a simple calculation, because the kidney receives blood to regulate the blood volume and composition, not for their own benefit.

Increased renal blood flow increases the glomerular filtration rate, which in turn must increase the rate of sodium reabsorption, increasing tissue oxygen consumption. Inability to increase delivery without increasing the demand may cause chronic hypoxia. And indeed recent studies using DW MRI and BOLD MRI have demonstrated renal parenchymal hypoxia of CKD patients with or without diabetes.

Chronic hypoxia is one of the major key insults affecting the diabetic kidney as hyperglycemia and hyperfiltration triggers a vicious circle between increasing oxygen delivery and increasing oxygen consumption that leads to more need for oxygen supply. Pseudohypoxia also exists due to hyperglycemia induced mitochondrial oxygen consumption. Hypoxia/pseudohypoxia contributes to the induction of TGF Beta1, MAPK, which have important role in these pathological mechanisms.

Dissociation between demand and delivery can only be achieved by increasing oxygen delivery using hyperbaric oxygen therapy.

Hyperbaric oxygen therapy (HBOT)

Hyperbaric oxygen therapy (HBOT) includes the inhalation of 100% oxygen at pressures exceeding 1 atmosphere absolute (ATA) in order to enhance the amount of oxygen dissolved in the body tissues. During HBOT treatment, the arterial O2 tension typically exceeds 2000 mmHg, and levels of 200-400 mmHg occur in tissues.

As explained in detail by Efrati and Ben-Jacob, the diverse and powerful innate repair mechanisms activated by HBOT are associated both with the elevated level of dissolved oxygen and with the elevated pressure.

Hyperbaric oxygen therapy has been used for years for the treatment of ischemic diabetic ulcers. The sharp increase in tissue oxygenation enables angiogenesis and regeneration.

The same effects on brain ischemic lesions have been comprehensively studied, reviling improved perfusion and function after a course of HBO treatment.

Breathing oxygen under hyperbaric conditions elevates the capillary dissolved oxygen partial pressure significantly, which enables maximal passive diffusion of oxygen from the capillary to the mitochondria in all tissues.

Hyperbaric oxygen upregulate the expression of hypoxia-inducible-factor-1alpha (HIF-1a).probably via sensation of relative decrease from hyperoxia to normoxia, which could be sensed as relative hypoxia. HIF-1a increases the transcriptional activity of VEGF and its mRNA stability, improves vascular permeability, and eliminates edema.

HBOT and stem cells:

HBOT induces stem cells mobilization from bone marrow. The number of circulating stem cells increases up to 3-8 times compared to pretreatment level . Mobilized stem cells have higher concentrations of an array of regulatory proteins such as hypoxia inducible factors, which in the murine model exhibit improved neovascularization.

Studies have shown that stem cells mobilized by HBOT home in on tissues that have suffered damage and signal a need for regeneration, such as in the case of diabetic chronic ulcers or radiation related injuries.

HBOT and the kidneys:

The effect of HBO on the diabetic kidney has never been studied in human. However few studies have analyzed it's effect in animal diabetes model. Hyperbaric oxygen therapy (HBOT) suppresses biomarkers of cell stress and kidney injury in diabetic mice. And the treatment was found to be safe for renal function in another study with rats.

The aim of the present study is to evaluate the effect of HBO on a wide range of kidney functions and markers in patients with diabetic nephropathy.

Methods

The study is as a prospective, controlled trial conducted in the Segol hyperbaric institute and the research unit of Assaf-Harofeh Medical Center. All patients will sign a written informed consent. The protocol was approved by Assaf-Harofeh institutional review board.

After signing an informed consent form, patients are invited for baseline evaluation. Analysis of urine, blood, pulse wave analysis and fMRI will be done at baseline, after the follow up period and after the treatment period are done, after which patients will be randomly assign to either follow up or HBOT treatment. The analysis listed above will be repeated by the end of the first period, and then patients will be cross over to either HBOT or follow up. The following HBOT protocol will be practiced: 60 daily sessions, 5 days/week, 120 minutes each, 100% oxygen at 2ATA.

ELIGIBILITY:
Inclusion Criteria:

* The participants are patients of age 18 years or older, who suffered DKD, defined as eGFR<60ml/min as estimated using MDRD formula, and albuminuria in the presence of diabetes. Diabetic retinopathy and without any alternative cause for their renal disease.

Exclusion Criteria:

* Exclusions criteria are chest pathology incompatible with HBOT, inner ear disease, claustrophobia. Smoking is not allowed during the study. Patients with uncontrolled diabetes HBA1C>7.5, recent AKI (3M) recent cardiovascular or cerebrovascular event (6M) or inability to hold the breath for 20-30 seconds are also excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
glomerular filtration rate | within a month after treatment
proteinuria | within a month after treatment

SECONDARY OUTCOMES:
renal blood flow (BOLD) | within a month after treatment
fibrosis (DWI MRI) | within a month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Keren Doenyas, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Dialysis Clinic in Asaf Harofhe Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No